CLINICAL TRIAL: NCT04030897
Title: Promoting Treatment Access Following Pediatric Primary Care Depression Screening: Evaluation of Web-based, Single-session Interventions for Parents and Youths
Brief Title: Promoting Treatment Access Following Pediatric Primary Care Depression Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2019-00241
Record Dates: First submitted 2019-07-20; First posted 2019-07-24 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Youths reporting elevated MD symptoms at a PC visit (N = 200) will be randomly assigned to one of two conditions (within a waitlist-control design): Information, Psychoeducation, and Referral (IPR; ie., usual care, or the "control") or IPR enhanced with youth- and parent-directed online SSIs (IPR+SSI), designed to reduce youth MD symptoms and improve parents' expectancies of mental health treatment, respectively.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participating youths and parents will be aware of whether they are receiving the online interventions immediately or after the 3-month follow-up period (i.e., whether they are in the 'intervention group' or the 'waitlist group'). However, participating families will be assigned to these conditions via an online survey, which they complete remotely, and condition assignments will be unknown to the research team and the youth's primary care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Programs + Information/Psychoeducation/Referral (IPR) (Active Comparator): Includes 2 online, one-session programs (one for youths; one for parents) and Primary Care-based IPR. The 30-min, self-administered YOUTH PROGRAM includes: An introduction to the brain and a lesson on neuroplasticity; Testimonials from older youths who describe their views that traits are malleable, due to the brain's plasticity; Further stories by older youths, describing times when they used "growth mindsets" to persevere during social/emotional setbacks; Study summaries noting how/why personality can change; And an exercise in which youths write notes to younger students, using scientific information to explain people's capacity for change. In the 15-min Qualtrics-based PARENT PROGRAM, parents read 2 scientific passages on (1) the notion that emotions are flexible in youth and adults, and (2) that failure promotes personal growth. After each passage, parents write a persuasive summary of its main arguments, directed to fellow parents who may benefit from the information.
  Interventions: Behavioral: Parent-Directed Online Single-Session Program; Behavioral: Youth-Directed Online Single-Session Program; Behavioral: Information/Psychoeducation/Referral
- Information/Psychoeducation/Referral (IPR; usual care control) (Placebo Comparator): Information, Psychoeducation and Referral (IPR) represents usual care in the Stony Brook University Hospital's Pediatric Primary Care Division. Families of a youth with elevated MD symptoms during a PC visit receive a folder containing informational materials about the nature of depression and referrals to providers in their area. All families in this study will receive PC-based IPR.
  Interventions: Behavioral: Information/Psychoeducation/Referral

INTERVENTIONS:
Behavioral: Parent-Directed Online Single-Session Program — Online, 15-minute self-administered program for parents
  Arms: Online Programs + Information/Psychoeducation/Referral (IPR)
Behavioral: Youth-Directed Online Single-Session Program — Online, 30 minute self-administered program for youths
  Other Names: Project Personality
  Arms: Online Programs + Information/Psychoeducation/Referral (IPR)
Behavioral: Information/Psychoeducation/Referral — Usual care at pediatric primary care clinics participating in this study

SUMMARY:
Major depression (MD) in youth is a serious psychiatric illness with extensive morbidity and mortality. The American Academy of Pediatrics recently released practice guidelines promoting primary care (PC)-based youth MD screening; however, even when diagnosed by PC providers, <50% of youth with MD access treatment. Thus, a need exists for interventions that are feasible for youths and parents to access and complete-and that may strengthen parents' likelihood of pursuing longer-term services. Single-session interventions (SSIs) may help forward these goals. SSIs include elements of comprehensive treatments, but their brevity makes them easier to disseminate at scale. Meta-analytic evidence suggests SSIs can reduce youth psychopathology, including self-administered (e.g., online) SSIs. One computer-based SSI, teaching growth mindset (GM; viewing personal traits as malleable), has reduced adolescent depressive symptoms in multiple RCTs; GM-SSIs have also improved parents' expectancies that psychotherapy could benefit their children's mental health. This project will test whether these online, youth- and parent-directed GM-SSIs-designed to reduce youth depressive symptoms and improve parents' mental health treatment expectancies, respectively-may increase mental health service access, reduce youth depressive symptoms, and relieve parental stress following PC-based youth MD screening. Youths reporting elevated MD symptoms at PC visits (N = 200) will receive either Information/Psychoeducation/Referral (IPR) or IPR plus parent- and youth-directed GM-SSIs (IPR+SSI). The investigators will examine whether IPR+SSI, versus IPR alone, increases MD service access; reduces parental stress; and reduces youth depressive symptoms across three months. Results may yield a disseminable model for promoting youth treatment access after PC-based depression screening.

ELIGIBILITY:
Inclusion Criteria:

* Youth is between the ages of 11 and 16, inclusive, at the time of study recruitment
* Youth reports a Pediatric Symptom Checklist 'Internalizing' score of 5 or higher (out of 10) at her/his most recent pediatric primary care visit at 1 of the 9 Stony Brook University-affiliated clinics participating in this study
* Parent and youth are comfortable with reading and writing in English
* Parent and youth are comfortable with online activity

Exclusion Criteria:

* Parent or youth is not comfortable reading and/or writing in English
* Parent or youth is not comfortable with online activity

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Mental Health Treatment-Seeking Behavior Checklist | Baseline to 3-month follow-up
  At baseline and 3-month follow-up, parents will indicate whether they have engaged in each of four treatment-seeking behaviors for their child: researched local mental healthcare providers/agencies for their child; contacted a mental healthcare provider or agency about treatment for their child; contacted child's school regarding mental health supports for their child; and scheduled an appointment OR placed child on a waiting-list with a mental healthcare provider/agency. Total number of treatment-seeking behaviors between baseline and 3-month follow-up may range from 0 to 4. Individual behaviors are self-reported by parents on as 'yes' or 'no' (noting whether they engaged in the behavior during the study period). At baseline, parents will report on whether they engaged in these behaviors 'since the child's last doctor's appointment.' At follow-up, parents will report whether they have engaged in these behaviors 'since their past survey, 3 months ago.'
Change in Children's Depression Inventory 2 - Youth Report Total Score | Baseline to 3-month follow-up.
  Change in youth reported depressive symptoms, total score derived from 28-item CDI-2. Scores range from 0-56, with higher scores indicating higher levels of depression.

SECONDARY OUTCOMES:
Change in Pediatric Symptom Checklist - Youth-Report Total score | Baseline to 3-month follow-up.
  Youth-report measure of overall youth psychopathology. Youth rate 35 items on a 0-2 scale reflecting internalizing, externalizing, and attention-related symptoms. Scores range from 0 - 70. Higher scores indicate higher overall symptom severity.
Change in Pediatric Symptom Checklist- Parent Report Total score | Baseline to 3-month follow-up.
  Youth-report measure of overall youth psychopathology. Youth rate 35 items on a 0-2 scale reflecting internalizing, externalizing, and attention-related symptoms. Scores range from 0 - 70. Higher scores indicate higher overall symptom severity.
Change in Pediatric Symptom Checklist- Youth Internalizing Score (parent report) | Baseline to 3-month follow-up.
  Parent-report measure of overall youth psychopathology. Parents rate 5 items on a 0-2 scale reflecting internalizing symptoms in their child. Scores range from 0-10. Higher scores indicate higher overall symptom severity.
Change in Beck Hopelessness Scale - 4 (Youth Report) | Baseline to immediate post-online-intervention (in active intervention group only) and 3-month follow-up (between groups).
  Respondents (youths) report agreement with 4 items indicating levels of hopelessness about the future. Higher summed scores reflect greater levels of hopelessness, and scores range from 0-12.
Change in Beck Hopelessness Scale - 4 (Parent Report) | Baseline to immediate post-online-intervention (in active intervention group only) and 3-month follow-up (between groups).
  Respondents (parents) report agreement with 4 items indicating levels of hopelessness about the future. Higher summed scores reflect greater levels of hopelessness, and scores range from 0-12.
Change in Brief Symptom Inventory - 18 | Baseline to 3-month follow-up
  The Brief Symptom Inventory-18 (BSI-18) assesses self reported parent psychopathology and distress. Adult respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale. The total sum score yields an additional total distress score (range: 0-72). Higher scores indicate higher levels of overall psychological distress.
Change in Barriers to Accessing Care Evaluation (BACE) | Baseline to 3-month follow-up
  Parents rate the 30 items on a 0-3 scale indicating the degree to which various beliefs, concerns, circumstances, and logistical difficulties have stopped, delayed or discouraged them from getting professional care for their child's mental health problem. Higher total scores indicate greater perceived barriers to care. Scores range from 0-90, with higher scores indicating more overall barriers to accessing mental health care for their child.
Change in Attitudes Toward Therapy Scale - Parent | Baseline to immediate post-online-intervention (in active intervention group only) and 3-month follow-up (between groups).
  One-item measure used to assess parents' perceptions that therapy/counseling would be useful in reducing their child's emotional or behavioral difficulties, rated on a 0-10 scale (total score range: 0-10). Higher scores indicate stronger beliefs that therapy may help reduce mental health problems, whereas lower scores indicate weaker beliefs that therapy may help reduce mental health problems.
Mental Health Treatment Access at 3-month follow-up | 3-month follow-up
  Parents will indicate (yes/no) whether their child has received (a) new and/or (b) continuing school-based, outpatient, or other mental health-related services since the child's recent PC appointment (at baseline) and since the baseline assessment (at 3-month follow-up).
Change in Perceived Stress Scale | Baseline to 3-month follow-up
  The PSS is a well-validated measure of the degree to which situations in one's life are appraised as stressful, unpredictable, and uncontrollable. Higher total scores indicate greater overall perceived stress. The scale includes 10 items rated on a 0-4 scales, and scores range from 0-40.
Change in Pediatric Symptom Checklist - Youth-Report Internalizing Score | Baseline to 3-month follow-up.
  Youth-report measure of youth depressive symptoms. Youth rate 5 items reflecting internalizing symptoms on a scale from 0-2. Total scores range from 0 to 10. Higher scores indicate higher internalizing symptom severity.
Change in Children's Depression Inventory 2 - Parent Report total score | Baseline to 3-month follow-up.
  Parent reported youth depressive symptoms, total score derived from 17-item parent-report version of CDI-2. Scores range from 0-54, and higher scores indicate greater youth depression severity.

OTHER OUTCOMES:
Change in implicit theories of emotion scale, parent-report | Baseline to immediate-post-online intervention (active intervention group only)
  This measure will be used as a manipulation check for parents assigned to the active intervention condition. Parents will be asked to report the degree to which they view emotions as malleable (versus immutable) at pre- and post-intervention using a previously validated, 4-item assessment of emotion mindsets in adults. Four items are rated using a 1-to-6 Likert scale. Higher mean scores on these items indicate a stronger fixed emotion mindset, a lower scores, a stronger growth emotion mindset (range: 1-).
Change in Implicit Theories of Personality Questionnaire, youth-report | Baseline to immediate-post-online intervention (active intervention group only)
  This measure will be used as a manipulation check for youths assigned to the active intervention condition. Respondents rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-6 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher mean scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset (range: 1-6).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level participant data will be made publicly available on Open Science Framework upon completion of the grant period (August 2021).
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and a statistical analysis plan have been uploaded with this pre-registration.
Access Criteria: Materials will be publicly available on clinicaltrials.gov. IPD will be made publicly available on Open Science Framework upon completion of the grant period (August 2021)

REFERENCES:
- [Derived] Schleider JL, Dobias M, Fassler J, Shroff A, Pati S. Promoting Treatment Access Following Pediatric Primary Care Depression Screening: Randomized Trial of Web-Based, Single-Session Interventions for Parents and Youths. J Am Acad Child Adolesc Psychiatry. 2020 Jun;59(6):770-773. doi: 10.1016/j.jaac.2020.01.025. Epub 2020 Apr 28. No abstract available. PMID 32666919

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT04030897/Prot_SAP_002.pdf